CLINICAL TRIAL: NCT01002781
Title: Efficacy and Safety of Tocilizumab (a Monoclonal Antibody to Receptor of IL-6) in the Treatment of Adult's Still Disease
Brief Title: Efficacy and Safety of Tocilizumab in Adult's Still Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Rambam Health Care Campus (Other); Assaf-Harofeh Medical Center (Other Government); Bnai Zion Medical Center (Other Government)
Responsible Party: Ori Elkayam, Israeli Society of Rheumatology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0452-09
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-09

CONDITIONS: Adult's Still Disease
Keywords: Tocilizumab Still
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab, IV, 8 mg/kg, every 2 weeks

SUMMARY:
Patients with adult's Still disease suffer from acute inflammatory symptoms such as fever, arthritis, rash, and acute phase response often requiring high dose corticosteroids. In view of several case reports which have shown dramatic improvement in patients treated with Tocilizumab and a phase 2 study of this drug in children with Still's disease, the objective of the current study is to assess the efficacy and safety of Tocilizumab in patients with adult's Still disease.

DETAILED DESCRIPTION:
This is a multicenter, open, study designed to investigate the effect of Tocilizumab, a monoclonal antibody to IL-6 receptor, on the management of active adult-onset Still's disease.

Standard medication of corticosteroid will be given to all patients at the discretion of the treating physician.

Visits will include : screening visit, week o, week 2 , and every 4 weeks after during 52 weeks After complying with the inclusion and exclusion criteria, patients will start treatment with Tocilizumab at a dosage of 8 mg/kg, every 2 weeks Patients will be assessed every visit for the presence of fever, tender and swollen joint, rash, dosage of corticosteroids and other DMARD's, CRP and ESR

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been diagnosed with adult-onset Still's disease according to the criteria of Yamaguchi (at least 5 criteria in total, including at least 2 major criteria), although these criteria do not have to be present at the time of inclusion in the study.

Major criteria are:Fever ≥39°C for at least 1 week,Arthralgia lasting at least 2 weeks,Maculo-papular, non-pruritic skin rash,Leucocytosis .≥10,000/mm³) including ≥80% neutrophils;Minor criteria are:Pharyngitis or sore throat,Lymphadenopathy or splenomegaly,Liver enzyme (transaminase) abnormalities,Negative for rheumatoid factor or antinuclear antibodies

* Patients aged >18
* Capable of signing informed consent

Exclusion Criteria:

* active infections (especially sepsis and Epstein-Barr virus),
* malignant disease (especially lymphomas),
* other autoimmune or inflammatory disease (especially polyarteritis nodosa)
* patients will be required to restrict other treatments for Still's disease to low-dose corticosteroids +/- non steroidal anti inflammatory drugs for at least the first 4 weeks of the study.
* pregnant or breast-feeding women
* women of childbearing potential unwilling to use adequate contraception and not become pregnant during the course of the study
* previous treatment with other biologic antirheumatic agents will require a washout period before inclusion
* history of listeriosis or latent or active tuberculosis
* persistent chronic or active recurring infection requiring treatment with antibiotics, antivirals, or antifungals within 4 weeks prior to the screening visit, or history of frequent recurrent infections unacceptable per investigator judgment.
* received administration of any live (attenuated) vaccine within 3 months prior to the inclusion visit
* known history of Human Immunodeficiency Virus antibody; and/or positive Hepatitis B surface antigen , and/or positive Hepatitis C antibody at the screening visit.
* history of recurrent herpes zoster.
* history of prior articular or prosthetic joint infection
* history of a hypersensitivity reaction, other than localised injection site reaction , to any biological molecule
* uncontrolled diabetes
* patients under dialysis
* presence of any of the following laboratory abnormalities at the screening visit: haemoglobin <8.5g/l, WBC <3000/μL, platelet count <150,000/μL, neutrophils <1500/μL
* AST or ALT >2 Upper limit and bilirubin >2 Upper limit

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
symptom-free or steroid-free remission at 52 weeks | 52 WEEKS

SECONDARY OUTCOMES:
fever, ACR20, inflammatory markers (e.g. CRP, ferritin), need for rescue medication (e.g. methotrexate, anti-TNF alpha) , adverse events | 52 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- Israel (4):
  - Bnei Tsion Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Tel Aviv Medical Center, Tel Aviv
  - Assaf Harofe Medical Center, Ẕerifin

REFERENCES:
- [Background] Yokota S, Imagawa T, Mori M, Miyamae T, Aihara Y, Takei S, Iwata N, Umebayashi H, Murata T, Miyoshi M, Tomiita M, Nishimoto N, Kishimoto T. Efficacy and safety of tocilizumab in patients with systemic-onset juvenile idiopathic arthritis: a randomised, double-blind, placebo-controlled, withdrawal phase III trial. Lancet. 2008 Mar 22;371(9617):998-1006. doi: 10.1016/S0140-6736(08)60454-7. PMID 18358927
- [Background] De Bandt M, Saint-Marcoux B. Tocilizumab for multirefractory adult-onset Still's disease. Ann Rheum Dis. 2009 Jan;68(1):153-4. doi: 10.1136/ard.2008.088179. No abstract available. PMID 19088261
- [Background] Iwamoto M, Nara H, Hirata D, Minota S, Nishimoto N, Yoshizaki K. Humanized monoclonal anti-interleukin-6 receptor antibody for treatment of intractable adult-onset Still's disease. Arthritis Rheum. 2002 Dec;46(12):3388-9. doi: 10.1002/art.10620. No abstract available. PMID 12483747